CLINICAL TRIAL: NCT01741558
Title: The Effects of mETHotrexate Therapy on ST Segment Elevation MYocardial InfarctionS: Randomized Double-blind, Placebo-controlled Trial (TETHYS Trial)
Brief Title: The Effects of mETHotrexate Therapy on ST Segment Elevation MYocardial InfarctionS (TETHYS Trial)
Acronym: TETHYS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Instituto de Cardiologia de Santa Catarina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UP 4747/12; CAAE 04482712.3.0000.5333 (Other: Plataforma Brasil)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Ischemia; Myocardial Infarction; Methotrexate; Inflammation; Anti-Inflammatory Agents; Inflammation Mediators
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia; Inflammation | interventions — Methotrexate; Riboflavin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methotrexate (Experimental): Established treatment associated with methotrexate
  Interventions: Drug: Methotrexate
- Placebo (Riboflavin) (Placebo Comparator): Established treatment associated with placebo (riboflavin sodium fosfate 0.1%). We use riboflavin in placebo group to remain the double-blind fashion: methotrexate has a yellow color and riboflavin in that concentration has the same color.
  Interventions: Drug: Riboflavin

INTERVENTIONS:
Drug: Methotrexate — The treatment group will receive a bolus dose of 0.05 mg/kg of methotrexate before primary angioplasty followed by 0.05 mg/kg per hour for 6 hours
  Other Names: Rheumatrex®; Trexall®; Amethopterin; MTX
  Arms: Methotrexate
Drug: Riboflavin — We use riboflavin in placebo group to remain the double-blind fashion: methotrexate has a yellow color and riboflavin in that concentration has the same color.
  Arms: Placebo (Riboflavin)

SUMMARY:
Experimental studies suggest that anti-inflammatory and immunomodulatory drugs could reduce the inflammatory profile in acute ischemic disease and reduce the area of ischemia. Methotrexate is a drug that has shown promise in ischemic disease in animal studies.

DETAILED DESCRIPTION:
Atherosclerosis and ischemic disease have clear association with inflammation. There is an anti-inflammatory action of methotrexate by increasing adenosine. Experimental studies demonstrate reduction of infarct induced in animals treated with methotrexate. We expect a reduction in the area under the curve of creatine kinase (CK), creatine kinase MB fraction (CK-MB) and Troponin I high sensitive, decreased levels of B-type natriuretic peptide (BNP) and improvement in left ventricular ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Chest pain suggestive of acute myocardial infarction initiated within 12 hours;
* Electrocardiogram with ST-segment elevation greater than or equal to 0.2 mV in at least 2 contiguous leads;
* Choice of primary angioplasty

Exclusion Criteria:

* Prior acute myocardial infarction;
* Prior heart failure;
* Angioplasty in the last 3 months;
* Cardiac arrest or cardiogenic shock;
* History of renal insufficiency (serum creatinine greater than 2.0 mg/dl);
* History of alcohol abuse (consumption equal to or greater than 20 drinks per week);
* Illicit drug use;
* Evidence of rheumatoid arthritis;
* Neoplasia;
* Infectious diseases;
* Prior anemia (hematocrit below 30%);
* Use of anti-inflammatory hormonal or non-hormonal last week;
* Xanthines excessive consumption (more than two and a half cups of coffee or two and a half mate gourds);
* Pregnancy;
* Disagreement with the term of consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve of creatine kinase | During 72 hours after the infarct
  The primary end point was the reduction of the size of the infarct as assessed by the area under the curve (AUC) (expressed in arbitrary units) for creatine kinase (CK) during 72 hours after the infarct

SECONDARY OUTCOMES:
Area under the curve for creatine kinase MB fraction and troponin I high sensitive | During 72 hours after the infarct
  The primary end point was the reduction of the size of the infarct as assessed by the area under the curve (AUC) (expressed in arbitrary units) for creatine kinase MB fraction(CK-MB) and Troponin I high sensitive during 72 hours after the infarct
Compare the peaks of CK, CK-MB and troponin I ultra-sensitive | During 72 hours after the infarct
  Compare the peaks of CK, CK-MB and troponin I ultra-sensitive
Compare the levels of high-sensitivity C-reactive protein at admission, after 72 hours and after 3 months | After 72 hours and after 3 months
  Compare the levels of high-sensitivity C-reactive at admission, after 72 hours and after 3 months
Compare the levels of erythrocyte sedimentation rate on admission and after 72 hours | On admission and after 72 hours
  Compare the levels of erythrocyte sedimentation rate on admission and after 72 hours
Compare B-type natriuretic peptide (BNP) levels on admission, after 72 hours and after 3 months | On admission, after 72 hours and after 3 months
  Compare B-type natriuretic peptide (BNP) levels on admission, after 72 hours and after 3 months
Compare the "TIMI frame count" of the culprit artery | On admission
  Compare the "TIMI frame count" of the culprit artery
Compare the Killip score on admission and after 72 hours | On admission and after 72 hours
  Compare the Killip score on admission and after 72 hours;
Assess ventricular ejection fraction with transthoracic echocardiography during the first 72 hours after 3 months | During the first 72 hours after 3 months
  Assess ventricular ejection fraction with transthoracic echocardiography during the first 72 hours after 3 months
Assess mortality at 3 months | At 3 months;
  Assess mortality at 3 months;
Evaluate reinfarction in 3 months | In 3 months
  Evaluate reinfarction in 3 months
Rate side effects | In 72 hours
  Evaluation in 72 hours the changes in the levels of hematocrit, hemoglobin, leukocytes and platelets, changes in the levels of serum glutamate oxaloacetate transaminase, serum glutamate pyruvate transaminase and prothrombin Time; changes in the levels of plasma creatinine, gastrointestinal effects (oral ulcers, diarrhea, nausea and vomiting), skin changes (rash, pruritus, and alopecia) and pulmonary effects (pneumonitis and pneumonia).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Moreira, MD. MSc., Study Chair — Instituto de Cardiologia do Rio Grande do Sul; Daniel M. Moreira, MD. MSc, Study Director — Instituto de Cardiologia do Rio Grande do Sul; Daniel M. Moreira, MD. MSc., Principal Investigator — Instituto de Cardiologia do Rio Grande do Sul; Carlos AM Gottschall, MD MSc PhD, Study Director — Instituto de Cardiologia do Rio Grande do Sul; Maria E. Lueneberg, MD., Study Director — Instituto de Cardiologia de Santa Catarina; Roberto L. da Silva, MD., Study Director — Instituto de Cardiologia de Santa Catarina; Tammuz Fattah, MD., Study Director — Instituto de Cardiologia de Santa Catarina
Locations (2):
- Brazil (2):
  - Instituto de Cardiologia do Rio Grande do Sul / Fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia de Santa Catarina, São José, Santa Catarina

REFERENCES:
- [Derived] Moreira DM, Lueneberg ME, da Silva RL, Fattah T, Gottschall CAM. MethotrexaTE THerapy in ST-Segment Elevation MYocardial InfarctionS: A Randomized Double-Blind, Placebo-Controlled Trial (TETHYS Trial). J Cardiovasc Pharmacol Ther. 2017 Nov;22(6):538-545. doi: 10.1177/1074248417699884. Epub 2017 Mar 22. PMID 28325070